CLINICAL TRIAL: NCT02467465
Title: Efficacy of Dry Needling in Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Miguel Suárez Varela, Physiotherapy degree, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Univ. Complutense de Madrid
Record Dates: First submitted 2015-05-27; First posted 2015-06-10 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-07

CONDITIONS: Fasciitis, Plantar
Keywords: Fasciosis plantar; physiotherapy; fascitis plantar; dry needling
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical therapy modalities (Experimental): Manual therapy techniques aimed to relaxed gastrocnemius and soleus muscles tone, movilizations, stretching and home exercises.
  Interventions: Other: Physical therapy modalities
- Invasive Physical therapy modalities (Experimental): Manual therapy techniques aimed to relaxed gastrocnemius and soleus muscles tone, movilizations, stretching and home exercises. Previously, DN will be applied in gastrocnemius and soleus muscles.
  Interventions: Other: Physical therapy modalities; Device: Invasive Physical therapy modalities

INTERVENTIONS:
Other: Physical therapy modalities — Massage, movilization of ankle dorsiflexion and improve flexibility with stretching of calf muscles.
Device: Invasive Physical therapy modalities — Dry needling added to massage, movilization of ankle dorsiflexion and improve flexibility with stretching of calf muscles.
  Arms: Invasive Physical therapy modalities

SUMMARY:
The plantar fasciitis (PF) is the most common cause of pain on the underside of the heel. About 10% to 20% of the population suffer once during their lifetime. PF concept began to describe at the end of XX century through the discovery of new clinical and histopathological signs of the plantar fascia. The difficulty of diagnosis, understanding and treatment of PF require us to develop new treatment avenues to improve the approach and the understanding of it. Dry needling (DN) as a treatment of myofascial pain syndrome (MPS) and myofascial trigger points (MTP) of muscle associated with the pathology, it may be a good treatment strategy, as demonstrated in the treatment of MPS in other body regions such as the neck, shoulder or the lumbar spine.

DETAILED DESCRIPTION:
Hypothesis:

Add dry needling to a physiotherapy intervention, increases the efficacy of treatment for plantar fasciosis.

Objectives:

General:

Test the efficacy of DN in addition to physiotherapy treatment includes: manual therapy and home exercises; directed to normalize muscle tone and inhibit MTP of the gastrocnemius and soleus muscles, in a group of patients who have been diagnosed with PF.

The variables to measure the efficacy are:

Pain assessment in the affected heel, by visual analog scale (VAS). Ultrasonographic assessment of the thickness of the plantar fascia affected, in longitudinal view, compared with the contralateral.

Goniometric assessment of joint range of ankle dorsiflexion, compared with the contralateral.

Specific:

Analyze the efficacy of the combination of DN treatment with manual therapy and home exercise, in patients who have been diagnosed with PF through monitoring and comparison between groups.

Methodology:

Type of study: clinical trial.

Sample:

It has been used sample size calculator GRANMO version 7.12, and accepting an alpha risk of 0.05 and a beta risk of 0.2, 15 subjects were required in the first group and 15 in the second to detect a difference equal to or greater than 0.6 units. It is assumed that the common standard deviation is 0.57. It has been estimated loss rate of 0%.

population: patients with a confirmed diagnosis of PF, who agree to participate in the study after signing the informed consent and carry out the selection criteria.

Sample:

It has been used sample size calculator GRANMO version 7.12, and accepting an alpha risk of 0.05 and a beta risk of 0.2, 15 subjects were required in the first group and 15 in the second to detect a difference equal to or greater than 0.6 units. It is assumed that the common standard deviation is 0.57. It has been estimated loss rate of 0%.

Selection criteria:

Ultrasonographic study in which a proximal thickened affected plantar fascia is observed greater than or equal to 4 mm.

Pain fell to the first steps in the morning. Pain with palpation at the insertion of the medial calcaneal tubercle, above 5, in a 10-point VAS.

Pathology time evolution of greater than or equal to 4 weeks. Age of patients over 18 years. Acceptance by the patient to participate in the study, having signed the informed consent.

Absence of neoplastic disease. Absence of neurological, sensory, orthopedic and / or surgical alterations. The patient is already doing treatment of physical medicine and rehabilitation. Be subjected to antiplatelet drug therapy. Fear of needles (needle phobia). Difficulty for the patient to understand the instructions to be followed during the study.

Methods of collecting information:

Personal data for each patient and relevant to the study, collected in a protocolized questionnaire, as well as an Excel sheet. All this in a personal history, encoded according to a table of alphanumeric equivalents, allowing subsequent statistical analysis with SPSS19.0 program.

Statistical method:

Initially, a descriptive statistical analysis will be conducted: qualitative variables were summarized by frequency distribution and quantitative by its average and standard deviation. Also it summarizes the information graphically using box plots, bar charts and pie charts.

Furthermore an inferential analysis using parametric or non-parametric techniques, particularly for the main objective analysis of variance was used in two groups (assuming a normal distribution for the variable response) U test or Mann-Whitney will be made in the case lack of normal. To study the response variables in each test group the Student t test or unimuestral averages Wilcoxon signed ranks for related samples was used.

For the analysis of qualitative variables the test of Chi-square test and the association between quantitative variables will be analyzed using the Pearson correlation coefficients and Spearman.

To test these significant differences in values of p <0.05 was assumed. Statistical analysis was performed using the statistical software SPSS v19.0

ELIGIBILITY:
Inclusion Criteria:

* Ultrasonographic study in which a proximal thickened affected plantar fascia is observed -greater than or equal to 4 mm.
* Pain fell to the first steps in the morning.
* Pain with palpation at the insertion of the medial calcaneal tubercle, above 5, in a 10-point VAS.
* Pathology time evolution of greater than or equal to 4 weeks.
* Age of patients over 18 years.
* Acceptance by the patient to participate in the study, having signed the informed consent.

Exclusion Criteria:

* Presence of neoplastic disease.
* Presence of neurological, sensory, orthopedic and / or surgical alterations.
* The patient is already doing treatment of physical medicine and rehabilitation.
* Be subjected to antiplatelet drug therapy.
* Fear of needles (needle phobia).
* Difficulty for the patient to understand the instructions to be followed during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suárez Miguel, Physician, Principal Investigator — Principal Investigator
Locations (1):
- Clínica Universitaria de Podología de la Universidad Complutense de Madrid, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Physical Therapy Modalities: Manual therapy techniques aimed to relaxed gastrocnemius and soleus muscles tone, movilizations, stretching and home exercises.
  Physical therapy modalities: Massage, movilization of ankle dorsiflexion and improve flexibility with stretching of calf muscles.
  Primary completion date is after January 2017.
- Invasive Physical Therapy Modalities: Manual therapy techniques aimed to relaxed gastrocnemius and soleus muscles tone, movilizations, stretching and home exercises. Previously, DN will be applied in gastrocnemius and soleus muscles.
  Invasive Physical therapy modalities: Dry needling added to massage, movilization of ankle dorsiflexion and improve flexibility with stretching of calf muscles.
  Primary completion date is after January 2017.
- Total: Total of all reporting groups
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.67 (11) | 49.47 (12.44) | 51.57 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  Spain | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Ultrasonographic Evaluation of the Thickness of the Affected Plantar Fascia, in Longitudinal View.
Description: Plantar fascia thickness in millimeters with ultrasonography at 0,5 centimeters from the calcaneo bone. Mean of 3 measures was taken.
Time Frame: 1 day.
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
millimeters | 5.3 [4.8 to 6.5] | 4.7 [4.3 to 5.5]

2. Primary Outcome: Ultrasonographic Evaluation of the Thickness of the Affected Plantar Fascia, in Longitudinal View.
Description: as for outcome 1
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
millimeters | 5.0 [4.3 to 5.8] | 4.2 [3.7 to 4.9]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.175, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Ultrasonographic Evaluation of the Thickness of the Affected Plantar Fascia, in Longitudinal View.
Description: as for outcome 1
Time Frame: 3 month
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
millimeters | 4.6 [4.1 to 5.8] | 4.0 [3.6 to 4.4]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.250, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Ultrasonographic Evaluation of the Thickness of the Affected Plantar Fascia, in Longitudinal View.
Description: as for outcome 1
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: millimeters
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
millimeters | 4.4 [4.0 to 5.9] | 3.9 [3.6 to 4.2]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.466, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Pain Assessment in the Affected Heel, by Visual Analog Scale.
Description: First step pain measured by Visual Analogue Scale, from 0 to 10 points, in the affected heel. In the Visual Analogue Scale, 0 represents the lowest score and 10 represents the highest score when the patient felt the maximum level of pain.
Time Frame: 1 day.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 8 [7 to 8] | 7 [5 to 8]

6. Secondary Outcome: Pain Assessment in the Affected Heel, by Visual Analog Scale.
Description: as for outcome 5
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 3 [2 to 6] | 2 [0 to 4]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.737, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Pain Assessment in the Affected Heel, by Visual Analog Scale.
Description: as for outcome 5
Time Frame: 3 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 2 [0 to 3] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.275, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Pain Assessment in the Affected Heel, by Visual Analog Scale.
Description: as for outcome 5
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.066, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Pain Assessment in the Affected Heel After Long Periods of Rest, by Visual Analog Scale.
Description: Pain after long periods of rest measured by Visual Analogue Scale, from 0 to 10 points, in the affected heel. In the Visual Analogue Scale, 0 represents the lowest score and 10 represents the highest score when the patient felt the maximum level of pain.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 7 [5 to 8] | 7 [5 to 8]

10. Secondary Outcome: Pain Assessment in the Affected Heel After Long Periods of Rest, by Visual Analog Scale.
Description: as for outcome 9
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 4 [2 to 5] | 4 [0 to 5]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.849, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Pain Assessment in the Affected Heel After Long Periods of Rest, by Visual Analog Scale.
Description: as for outcome 9
Time Frame: 3 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 0 [0 to 2] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.425, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Pain Assessment in the Affected Heel After Long Periods of Rest, by Visual Analog Scale.
Description: as for outcome 9
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
units on a scale | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.487, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Extended.
Description: Range of motion of ankle dorsiflexion with knee extended measured in grades using a goniometer. There is not exist minimum and maximum scores for the goniometric assessment, because the limits of the range of motion depends on the joint mobility, then, for this measure, higher values are better results than lower values. Clinically, it means that one patient with 100 degrees of range of motion has more mobility than another with 90 degrees.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 95 [92 to 100] | 99 [92 to 105]

14. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Extended.
Description: Range of motion of ankle dorsiflexion with knee extended measured in grades using a goniometer. There is not exist minimum and maximum scores for the goniometric assessment, because the limits of the range of motion depends on the joint mobility, then, for this measure, higher values are better results than lower values.Clinically, it means that one patient with 100 degrees of range of motion has more mobility than another with 90 degrees.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 101 [96 to 105] | 104 [100 to 108]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.651, t-test, 1 sided

15. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Extened.
Description: as for outcome 13
Time Frame: 3 month
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 100 [98 to 109] | 104 [98 to 109]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.387, t-test, 1 sided

16. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Extended.
Description: as for outcome 13
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 104 [101 to 110] | 108 [100 to 112]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.755, t-test, 1 sided

17. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Flexed.
Description: Range of motion of ankle dorsiflexion with knee flexed 90º measured in grades using a goniometer. There is not exist minimum and maximum scores for the goniometric assessment, because the limits of the range of motion depends on the joint mobility, then, for this measure, higher values are better results than lower values. Clinically, it means that one patient with 100 degrees of range of motion has more mobility than another with 90 degrees.
Time Frame: 1 day
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 104 [101 to 108] | 109 [100 to 112]

18. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Flexed.
Description: as for outcome 17
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 108 [105 to 115] | 110 [100 to 113]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.032, t-test, 1 sided

19. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Flexed.
Description: as for outcome 17
Time Frame: 3 month
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 109 [106 to 113] | 110 [106 to 111]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.058, t-test, 1 sided

20. Secondary Outcome: Goniometric Assessment of Joint Range of Motion Ankle Dorsiflexion With Knee Flexed.
Description: as for outcome 17
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
Number analyzed (Participants) | 15 | 15
degrees | 110 [105 to 114] | 110 [106 to 115]
Statistical Analysis 1: Comparison: Physical Therapy Modalities vs Invasive Physical Therapy Modalities; Test type: Superiority; p = 0.279, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Physical Therapy Modalities | Invasive Physical Therapy Modalities
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Statistical Analysis Plan (2014-04-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02467465/SAP_000.pdf
  • Study Protocol (2014-04-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02467465/Prot_001.pdf
  • Informed Consent Form (2014-07-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT02467465/ICF_002.pdf